CLINICAL TRIAL: NCT06646185
Title: IMVAHA: Improving Menstrual and VAginal Health for All
Brief Title: Improving Menstrual and VAginal Health for All
Acronym: IMVAHA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: Universidad Nacional de la Amazonia Peruana (Unknown); Universidad Peruana Cayetano Heredia (Other); Centre de Recherche sur les Maladies Emergentes et Re-Emergentes (Unknown); Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Sonja Merten, Head of Unit Society, Gender and Health, Swiss Tropical & Public Health Institute
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2023-30
Record Dates: First submitted 2024-09-24; First posted 2024-10-17 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Effects of Menstrual Products on the Vaginal Microbiome
Keywords: vaginal microbiome; menstruation; crossover study; menstrual products
MeSH Terms: interventions — Menstrual Hygiene Products

STUDY DESIGN:
Intervention Model Description: A three-period crossover trial will study the effects of short-term use of 3 menstrual products (menstrual pad, tampon, menstrual cup) on the bacterial composition of the vaginal microbiome in three countries (Peru, Cameroon, and Switzerland). Each crossover period consists of two menstrual cycles, thus resulting in a 6-month trial. Participants will be randomly assigned to one of 6 exposure sequences (different order of products per sequence); in each sequence, participants will adopt each menstrual product for 2 menstrual cycles. Participants will provide vaginal microbiome samples via self-sample swabs at 3 points during each menstrual cycle. Given the crossover design of the study, there is not a dedicated control group. No wash-out period is included because participants can not stop the use of menstrual products to manage their menstruation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- TamponCupPad (Other): Participants will adopt tampons during the first two menstrual cycles (first period of the trial), followed by adoption of cups during the next two menstrual cycles (second period), and lastly menstrual pads for the next two menstrual cycles (third crossover period).
  Interventions: Other: Menstrual Pads; Other: Menstrual Cups; Other: Tampons
- TamponPadCup (Other): Participants will adopt tampons during the first two menstrual cycles (first period of the trial), followed by adoption of pads during the next two menstrual cycles (second period), and lastly menstrual cups for the next two menstrual cycles (third crossover period).
  Interventions: Other: Menstrual Pads; Other: Menstrual Cups; Other: Tampons
- CupTamponPad (Other): Participants will adopt menstrual cups during the first two menstrual cycles (first period of the trial), followed by adoption of tampons during the next two menstrual cycles (second period), and lastly menstrual pads for the next two menstrual cycles (third crossover period).
  Interventions: Other: Menstrual Pads; Other: Menstrual Cups; Other: Tampons
- CupPadTampon (Other): Participants will adopt menstrual cups during the first two menstrual cycles (first period of the trial), followed by adoption of menstrual pads during the next two menstrual cycles (second period), and lastly tampons for the next two menstrual cycles (third crossover period).
  Interventions: Other: Menstrual Pads; Other: Menstrual Cups; Other: Tampons
- PadTamponCup (Other): Participants will adopt menstrual pads during the first two menstrual cycles (first period of the trial), followed by adoption of tampons during the next two menstrual cycles (second period), and lastly menstrual cups for the next two menstrual cycles (third crossover period).
  Interventions: Other: Menstrual Pads; Other: Menstrual Cups; Other: Tampons
- PadCupTampon (Other): Participants will adopt menstrual pads during the first two menstrual cycles (first period of the trial), followed by adoption of menstrual cups during the next two menstrual cycles (second period), and lastly tampons for the next two menstrual cycles (third crossover period).
  Interventions: Other: Menstrual Pads; Other: Menstrual Cups; Other: Tampons

INTERVENTIONS:
Other: Menstrual Pads — Participants adopt menstrual pads to manage their menstruation during 2 menstrual cycles. For each menstrual cycle, participants will provide vaginal microbiome samples via self-sampled swabs at 3 points.
Other: Menstrual Cups — Participants adopt menstrual cups to manage their menstruation during 2 menstrual cycles. For each menstrual cycle, participants will provide vaginal microbiome samples via self-sampled swabs at 3 points.
Other: Tampons — Participants adopt tampons to manage their menstruation during 2 menstrual cycles. For each menstrual cycle, participants will provide vaginal microbiome samples via self-sampled swabs at 3 points.

SUMMARY:
A three-period crossover trial will study the effects of short-term use of 3 menstrual products (menstrual pad, tampon, menstrual cup) on the bacterial composition of the vaginal microbiome in three countries (Peru, Cameroon, and Switzerland). Each crossover period consists of two menstrual cycles, thus resulting in a 6-month trial. Participants will be randomly assigned to one of 6 exposure sequences (different order of products per sequence); in each sequence, participants will adopt each menstrual product for 2 menstrual cycles. Participants will provide vaginal microbiome samples via self-sample swabs at 3 points during each menstrual cycle. Given the crossover design of the study, there is not a dedicated control group.

DETAILED DESCRIPTION:
In three countries, the investigators will follow a randomized crossover design to study the effects of menstrual products on the vaginal microbiome composition and diversity. Eligible participants who are willing to adopt pads, tampons and menstrual cups to manage their menstruation, and for which baseline composition of their vaginal microbiomes is determined through DNA sequencing of the 16s rRNA gene will enter a three-period crossover trial. Each period of the trial will consist of two menstrual cycles, thus resulting in a 6-month trial. Participants will be randomly assigned to one of six different exposure sequences of menstrual products, as follows:

i) Tampon, Cup, Pad ii) Tampon, Pad, Cup iii) Cup, Tampon, Pad iv) Cup, Pad, Tampon v) Pad, Tampon, Cup vi) Pad, Cup, Tampon

In group "i)", participants will adopt tampons during the first two menstrual cycles (first period of the trial), followed by the adoption of cups during the next two menstrual cycles (second period), and lastly menstrual pads for the next two menstrual cycles (third crossover period). In groups ii) to vi) following the same design but in different sequences. Self-sampling kits will be provided during six consecutive menstrual cycles, a few days before the start of menses. Each kit will contain swabs for three self-sampling points during the menstrual cycle and the corresponding menstrual products.

ELIGIBILITY:
Inclusion Criteria:

* able to provide informed consent;
* aged 18-35;
* residing in the recruitment region and expecting to reside in the same region for at least six months following recruitment (Yaoundé/ Gounougou, Cameroon; Loreto/Lima/Maynas provinces, Peru; or Basel-Landschaft and Basel-Stadt cantons, Switzerland);
* are native speakers or are able to read and understand one of the following languages in each respective country (German, French, Italian, English or Spanish in Switzerland; French or English in Cameroon; Spanish in Peru);
* had menstrual cycles of 21-35 days for at least the last 4 months;
* had menses which lasted at least 3 days for at least the last 4 months.

Exclusion criteria:

* experienced a menstrual abnormality with any of the menstrual cycles in the last 4 months (such as oligomenorrhea or amenorrhea, or bleed more than 7 days a month);
* are pregnant or actively trying to become pregnant;
* are breastfeeding;
* used antibiotics and/or vaginal antifungals in the last 30 days prior to recruitment;
* had a vaginal birth in the last 6 months;
* vaginal surgery, perineal surgery, uterine surgery, miscarriage or abortion in the last 6 months;
* history of Toxic Shock Syndrome ;
* positive to detection of the toxic shock syndrome toxin-1 gen (tst) using Polymerase Chain Reaction (PCR);
* Intrauterine device in situ;
* under medication (treatment against infectious or chronic disease) at the time of recruitment or during the 3 weeks prior to recruitment;
* clinical symptoms of vaginal infection;
* smoker.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Log-ratio of Dialister to Lactobacillus crispatus relative abundances in vaginal swabs (continuous variable) | Monthly, after menstruation ends, through study completion, an average of 6 months.
  The abundances of each bacterial taxa are estimated from the DNA amplification and sequencing of amplicons from the 16S rRNA gene.

SECONDARY OUTCOMES:
Log-ratio of Bifidobacterium vaginalis to Lactobacillus relative abundances in vaginal swabs (continuous variable) | Monthly, after menstruation ends, through study completion, an average of 6 months.
  The abundances of each bacterial taxa are estimated from the DNA amplification and sequencing of amplicons from the 16S rRNA gene.
Log-ratio of Prevotella to Lactobacillus relative abundances in vaginal swabs (continuous variable) | Monthly, after menstruation ends, through study completion, an average of 6 months.
  The abundances of each bacterial taxa are estimated from the DNA amplification and sequencing of amplicons from the 16S rRNA gene.
Dominant taxon in vaginal swabs (categorical variable) | Monthly, after menstruation ends, through study completion, an average of 6 months.
  The dominant taxon in a vaginal swab is defined as the most abundant taxon found with a relative abundance of at least 30% of the total bacterial DNA sequences found in the sample.
Community state type in vaginal swabs (categorical variable) | Monthly, after menstruation ends, through study completion, an average of 6 months.
  The community state type in a vaginal swab is defined using the VALENCIA algorithm as described in this article: France, M.T., Ma, B., Gajer, P. et al. VALENCIA: a nearest centroid classification method for vaginal microbial communities based on composition. Microbiome 8, 166 (2020). https://doi.org/10.1186/s40168-020-00934-6
Total bacterial load in vaginal swabs (continuous variable) | Monthly, after menstruation ends, through study completion, an average of 6 months.
  Indirectly estimated with qPCR of the 16S rRNA gene
Self-reported vaginal complaints (discrete variable) | Monthly, from enrollment until study completion, an average of 6 months.
  Self-reported through follow up surveys along the six-month trial
Vaginal pH (ordinal variable) | Monthly, after menstruation ends, through study completion, an average of 6 months.
  Measured with a vaginal swab and a fixed indicator (3.6 - 6.1), just after menstruation ends.
Alpha diversity (continuous variable) | Monthly, after menstruation ends, through study completion, an average of 6 months.
  Alpha diversity indices (e.g., Shannon, Simpson) are estimated for each vaginal swab sample to quantify microbial richness and evenness.
Log-ratio of Gardnerella module to L. crispatus module relative abundances (continuous variable) | Monthly, after menstruation ends, through study completion, an average of 6 months.
  The abundances of each bacterial module are estimated from the DNA amplification and sequencing of amplicons from the 16S rRNA gene.
Log-ratio of Prevotella module to L. crispatus module relative abundances (continuous variable) | Monthly, after menstruation ends, through study completion, an average of 6 months.
  The abundances of each bacterial module are estimated from the DNA amplification and sequencing of amplicons from the 16S rRNA gene.
molBV score (discrete variable) | Monthly, after menstruation ends, through study completion, an average of 6 months.
  The molBV score in a vaginal swab is defined and derived as described in this article: Usyk, M., Schlecht, N.F., Pickering, S. et al. molBV reveals immune landscape of bacterial vaginosis and predicts human papillomavirus infection natural history. Nat Commun 13, 233 (2022). https://doi.org/10.1038/s41467-021-27628-3.

CONTACTS AND LOCATIONS:
Overall Officials: Sonja Merten, PhD, Principal Investigator — Swiss Tropical & Public Health Institute
Locations (3):
- Centre de Recherche sur les Maladies Emergentes et Re-Emergentes, Yaoundé, Yaoundé, Cameroon
- Universidad Nacional de la Amazonia Peruana, Iquitos, Iquitos, Peru
- Swiss Tropical and Public Health Institute, Allschwil, Allschwil, Switzerland

IPD SHARING:
Plan to Share IPD: No